CLINICAL TRIAL: NCT00125827
Title: A Phase I Dose Escalation and Pharmacokinetic Study of Oral Clofarabine Administered Daily for 5 Days in Adult Patients With Refractory Solid Tumors
Brief Title: Study of Oral Clofarabine Administered Daily for 5 Days in Adult Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO152
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Solid Tumors
Keywords: CLO152; Clolar
MeSH Terms: interventions — Clofarabine; Dosage Forms

ARMS (1):
- 1 (Experimental): Single-arm, dose escalation
  Interventions: Drug: clofarabine (oral formulation)

INTERVENTIONS:
Drug: clofarabine (oral formulation) — Cohorts of 3 patients each were to receive oral clofarabine administered daily for 5 days followed by 23 days of rest (1 cycle) and repeated every 28 days depending on toxicity and response. The starting dose of clofarabine was to be 1 mg/m2/day with subsequent dose escalation to occur in increments of 50% for the first 5 dose levels (1.5, 2.25, 3.5, and 5.0 mg/m2/day) and in increments of 25% thereafter until the MTD/RP2D was determined.

SUMMARY:
Clofarabine (injection) is approved by the Food and Drug Administration (FDA) for the treatment of pediatric patients 1 to 21 years old with relapsed acute lymphoblastic leukemia (ALL) who have had at least 2 prior treatment regimens.

This is a research study of clofarabine that will be given to patients (orally) with advanced cancerous tumors or cancerous tumors that have spread in which standard drugs are no longer effective or no reliable effective treatment is available.

The purpose of this study is to find the answers to the following research questions:

1. What is the largest dose of oral clofarabine that can be safely given daily for 5 days followed by 23 days of rest and repeated every 28 days?
2. What are the side effects of clofarabine when given on this schedule?
3. How much oral clofarabine is in the blood at specific times after administration and how does the body get rid of the drug?
4. Will oral clofarabine help treat solid tumor cancer?

ELIGIBILITY:
Inclusion Criteria:

* Have a pathologically confirmed diagnosis of a solid tumor malignancy that is refractory to conventional therapy or for which no therapy exists. Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Be greater than or equal to 18 years old.
* Must not be eligible for therapy of higher curative potential. (NB: Where an alternative therapy has been shown to prolong survival in an analogous population, that therapy will be offered to the patient prior to discussing this study.)
* Have a Karnofsky Performance Status (KPS) of greater than or equal to 70.
* Have an estimated life expectancy of greater than or equal to 12 weeks.
* Be male or a non-pregnant, non-lactating female. Patients who are fertile must agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy.
* Have a negative serum or urine pregnancy test within 10 days of study treatment (if patient is a female of childbearing potential).
* Sign a written informed consent form.
* Have adequate organ function as indicated by the following laboratory values, obtained within 2 weeks prior to registration: A. ANC: greater than or equal to 1.5 × 10 ^9th/L; B. Platelets: greater than or equal to 100 × 10 ^9th/L; C.Serum bilirubin: less than 2.0 mg/dL; D. AST and ALT: less than 3 x ULN* without liver involvement OR less than 5 x ULN with liver involvement; E. Serum creatinine: less than or equal to 2.0 mg/dL. NOTE: ULN = Institutional Upper Limit of Normal.

Exclusion Criteria:

* Have received previous treatment with clofarabine.
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Are pregnant or lactating.
* Have a psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
* Have received any chemotherapy, major surgery, or irradiation, whether conventional or investigational, 28 days before treatment in this study (42 days for mitomycin-C or nitrosourea).
* Have not recovered from acute toxicities of all previous therapy prior to enrollment.
* Have any other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study (eg, uncontrolled severe insulin-dependent diabetes, uncontrolled hypertension, transient ischemic attacks, uncontrolled symptomatic coronary artery disease, etc). Patients with abnormal cardiac function who are in consideration for study participation should be discussed with the Medical Monitor prior to enrollment.
* Have received prior radiation therapy to greater than or equal to 25% of the bone marrow (eg, no whole pelvic irradiation is allowed) and have not recovered from the acute side effects of radiotherapy.
* Have symptomatic or untreated central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-10; Primary Completion 2004-10 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD)/recommended phase II dose (RP2D) and dose limiting toxicity (DLT) of oral clofarabine when administered once daily for 5 days every 28 days to adult patients with locally advanced or metastatic solid tumors | Length of Study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Tyler Cancer Institute, Tyler, Texas
  - Cancer Care Northwest, Spokane, Washington